CLINICAL TRIAL: NCT07025772
Title: Approach Bias Retraining to Augment Long-Term Smoking Cessation Among a Diverse Sample
Brief Title: Shaping Habitual Impulses For a Tobacco-free Style
Acronym: SHIFTS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Lorra Garey, Research Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005124; RP250418 (Other Grant/Funding Number: Cancer Prevention and Research Institute of Texas)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: ST+ABR; ST+SHAM; ST-only
Keywords: Approach bias retraining; smoking cessation; cognitive retraining
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ST+ABR (Experimental): ST+ABR is the combination of standard treatment (cognitive behavioral therapy [CBT]+ nicotine replacement therapy [NRT]) for smoking cessation based on the most recent clinical practice guideline from the U.S. Department of Health and Human Services, Treating Tobacco Use And Dependence and computerized Approach Bias Retraining (ABR) for smoking cessation.
  Interventions: Behavioral: ST+ABR
- ST+Sham (Sham Comparator): ST+Sham is the combination of standard treatment (CBT+NRT) for smoking cessation based on the most recent clinical practice guideline from the U.S. Department of Health and Human Services, Treating Tobacco Use And Dependence and computerized Sham (Control) training.
  Interventions: Behavioral: ST+Sham
- ST Only (Other): ST Only will consist of standard treatment (CBT+NRT) for smoking cessation, based on the most recent clinical practice guideline from the U.S. Department of Health and Human Services, Treating Tobacco Use And Dependence.
  Interventions: Behavioral: ST Only

INTERVENTIONS:
Behavioral: ST+ABR — ST+ABR participants will complete seven weekly sessions of 15 minutes of computerized training (ABR), followed by a 45-minute session of standard smoking cessation treatment (CBT+NRT). Participants will be instructed to pull or push a joystick depending on the tilt, which will be positive-related or smoking-related images.
  Arms: ST+ABR
Behavioral: ST+Sham — ST+Sham participants will complete seven weekly sessions of 15 minute computerized control sessions (AAT), followed by a 45-minute session of standard smoking cessation treatment (CBT+NRT). Participants will be instructed to pull or push a joystick depending on the tilt, which will be positive-related or smoking-related images.
  Arms: ST+Sham
Behavioral: ST Only — ST Only will consist of 7 weekly 45-minute sessions of standard treatment (CBT+NRT) for smoking cessation.
  Arms: ST Only

SUMMARY:
The present investigation aims to assess the efficacy of an innovative and novel smoking cessation intervention that integrates approach bias retraining (ABR) and standard smoking cessation treatment (ST). Participants will be randomized to either: (1) standard smoking cessation treatment and approach bias retraining (ST+ABR); (2) ST+Sham; or (3) ST-only.

DETAILED DESCRIPTION:
The study employs a randomized controlled design to follow 300 individuals who smoke cigarettes as they engage in a smoking quit attempt following standard smoking cessation treatment (ST). Participants will be randomized to one of three conditions: (1) ST+ABR; (2) ST+Sham; or (3) ST-only. Participants will complete a self-screener, baseline appointment, 7 weeks of smoking cessation treatment, combined with approach bias retraining (if applicable) in the laboratory (with the quit day scheduled for the 6th session), 2x daily ecological momentary assessments (EMAs) for 4-weeks following their quit day, and 1-, 3-, and 6-month follow-ups in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

At least 18 years of age Ability to speak English fluently Ability to write in English fluently Smoke at least 5 cigarettes daily on average Smoke at least 5 cigarettes daily on average for the past year Motivated to quit smoking (≥ 5 on a 10-point scale) Willing to attend in-person visits Provide written informed consent, accepting study inclusion criteria and the randomized group assignment English literacy of 6th grade or higher, as indicated by a score of 4 or greater on the Rapid Estimate of Adult Literacy in Medicine-Short Form (REALM-SF) Biochemical verification of smoking status with expired carbon monoxide (CO) levels of >4 parts per million (PPM)

Exclusion Criteria:

Having used an e-cigarette in the past 3 months Having initiated any mental health therapy or pharmacotherapy within the past 3 months Being currently in therapy for substance abuse (including nicotine dependence) Currently using any NRT or psychotherapy products for nicotine cessation Currently using Bupropion as a smoking cessation aid and antidepressant Currently pregnant or planning to become pregnant Having high blood pressure that is not under control Having a heart attack within the past 2 weeks Having Visual impairments Hand-motoric impairments Currently suicidal or high suicide risk or current or past psychotic disorders of any type, bipolar disorder, schizophrenia or schizoaffective disorder, anorexia, bulimia Cognitive impairment, verified via a score of > 8 on the Six-Item Cognitive Impairment Test (6-CIT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
7-day Biochemically Verified Point Prevalence Abstinence (PPA) | [Time Frame: Baseline appointment through the 6-month follow-up, inclusive of every assessment (daily 2x EMAs for 4 weeks; 1-, 3-, and 6-month follow-ups)]
  PPA will be defined as no cigarette smoking within the past 7 days of assessments, and will be biochemically verified via assessment of expired carbon monoxide (<= 4ppm).
Prolonged Abstinence (PA) | [Time Frame: Baseline appointment through the 6-month follow-up, inclusive of every assessment]
  Participants will self report their abstinence by reporting whether or not they have smoked since their quit date.

CONTACTS AND LOCATIONS:
Locations (1):
- RESTORE Laboratory: Research on Emotion, Substance Use Treatment Outcomes, Rehabilitation, and Empowerment, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No